CLINICAL TRIAL: NCT03131102
Title: Association of Perioperative Early Tiredness (Acute Fatigue) With Hemodynamic, Immunologic, Endothelial, Metabolic, Gastrointestinal Measures and Complications in Patients With Epithelial Ovarian Cancer
Brief Title: Perioperative Early Tiredness (Acute Fatigue) in Patients With Epithelial Ovarian Cancer
Acronym: PERISCOPE
Status: Completed | Type: Observational
Sponsor: Aarne Feldheiser (Other)
Collaborators: Experimental & Clinical Research Center Berlin (Unknown); German Institute of Human Nutrition (Other); Humboldt-Universität zu Berlin (Other); Technische Universität Berlin (Other)
Responsible Party: Sponsor-Investigator, Aarne Feldheiser, Consultant, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Other Study IDs: PERISCOPE
Record Dates: First submitted 2017-03-27; First posted 2017-04-27 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Perioperative Early Tiredness (Acute Fatigue); Electrical Cardiometry; Biosignals; Mitochondrial Dysfunction; Nutrition
MeSH Terms: conditions — Mitochondrial Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Muscle biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with epithelial ovarian cancer (EOC): Patients undergoing cytoreductive surgery due to epithelial ovarian cancer
- Subgroup - Metabolomics in EOC patients without ascites: In a subgroup (n=10), patients without preoperative ascites will undergo extended metabolic measures to investigate mitochondrial dysfunction during the preoperative period.
- Subgroup - Metabolomics in EOC patients with ascites >500ml: In a subgroup (n=10), patients with preoperative ascites >500ml will undergo extended metabolic measures to investigate mitochondrial dysfunction during the preoperative period.

SUMMARY:
In surgical patients early risk prediction of postoperative complications and organ dysfunctions is still an important clinical challenge whereas appropriate risk predictors are still missing. In this regard, fatigue is a complex phenomenon, is affected by many factors and has been shown to be associated with delayed return to normal activity after surgery. The investigators hypothesize that early tiredness (acute fatigue) assessed shortly after surgery is associated to postoperative complications and organ dysfunctions and might be used for risk stratification. Therefore, in this prospective, observational study the investigators introduce and evaluate a newly developed score to assess early fatigue during the perioperative period ("Acute Fatigue Score", AFS).

The AFS and the Identity-Consequence Fatigue Scala will be used to assess early fatigue and perioperative time courses and inter-rater-variability will be evaluated. The rating of these two fatigue scores will be evaluated regarding the association with hemodynamic, immunologic, endothelial, metabolic, gastrointestinal measures as well as organ dysfunction and complications after surgery.

Furthermore, hemodynamic, immunologic, endothelial, metabolic and gastrointestinal measures are investigated with respect to the intraoperative course and postoperative organ dysfunction and complications. In a subgroup of patients, patients will undergo specialized metabolic measures to investigate mitochondrial dysfunction during the perioperative period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epithelial ovarian cancer scheduled for cytoreductive surgery at the Department of Gynecology at Campus Virchow - Klinikum, Charité - University Berlin
* Offered patient information and written informed consent

Exclusion Criteria:

* Patients aged less than 18 years
* Persons without the capacity to consent
* Inability of German language use
* Lacking willingness to save and hand out data within the study
* Accommodation in an institution due to an official or judicial order
* (Unclear) history of alcohol or substances disabuse
* Coworker of the Charité
* Known Myopathy
* Neurological or psychiatric disease at the beginning of hospitalization
* CHF (congestive heart failure) according to (New York Heart Association) classification - NYHA class IV at the beginning of hospitalization
* American Society of Anesthesiologists (ASA) classification greater than IV
* Renal insufficiency (dependency of haemodialysis) at the beginning of hospitalization
* Pulmonary oedema in thorax x-ray at the beginning of hospitalization
* History of intracranial hemorrhage within one year before participation in the study
* Conditions following venous thrombosis within the last three years before study inclusion
* Known allergies or hypersensitivity on colloidal, starch or gelatine infusion solutions
* Diabetes mellitus with signs of severe neuropathy
* Known atrial fibrillation
* Participation in an interventional clinical trial during the study period; exception: assignment to adjuvant therapy study during this study is allowed.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with epithelial ovarian cancer undergoing cytoreductive surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2017-08-29 (Actual); Primary Completion 2018-10-09 (Actual); Study Completion 2018-10-09 (Actual)

PRIMARY OUTCOMES:
Acute Fatigue Score (AFS) | 1 hour after the end of anaesthesia
  Rating of the AFS

SECONDARY OUTCOMES:
Acute Fatigue Score (AFS) | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before and after the first cycle of chemotherapy (an average of four to six weeks)
  Perioperative time course of the ratings of AFS
Inter-Rater Variability of Acute Fatigue Score (AFS) | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before and after the first cycle of chemotherapy (an average of four to six weeks)
  The scores will be assessed by two observers and the variability determined
Identity-Consequence Fatigue Scala (ICFS) | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before and after the first cycle of chemotherapy (an average of four to six weeks)
  Previously published score to measure tiredness
Hemodynamic variables and catecholamine administration | Up to the fifth postoperative day
  Hemodynamic variables are assessed by the anesthesia monitor
Hemodynamic variables obtained by Electrical Cardiometry (EC) | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before, during and after the first cycle of chemotherapy (an average of four to six weeks)
  EC is a method of bioimpedance
Hemodynamic shock indices calculated from Electrical Cardiometry (EC) | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before, during and after the first cycle of chemotherapy (an average of four to six weeks)
  EC is a method of bioimpedance
Heart rate variability, cardiorespiratory coupling, pulse wave velocity and new markers calculated from raw biosignals | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before, during and after the first cycle of chemotherapy (an average of four to six weeks)
  Bioelectrical signals to assess the interaction of the cardiac and pulmonary rhythms
Metabolomics/Proteomics | Up to the first postoperative day
  Metabolomic, proteomic, immunological, endothelial and inflammatory markers obtained by intramuscular microdialysis
Mitochondrial respiratory chain activities | Up to the first postoperative day
  Respiratory chain activities are assessed in muscle biopsies using high-resolution respirometry
Nutrition associated antibodies and deficiency states of vitamins and trace elements | Up to the fifth postoperative day
  Biochemical parameters of nutrition states and immunological marker of alimentary components are determined
Blood loss | Up to the fifth postoperative day
  Perioperative blood loss characteristics
Body temperature | Up to the first postoperative day
  Body temperature will be assessed continuously and discontinuously
Fluid balances | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before, during and after the first cycle of chemotherapy (an average of four to six weeks)
  The balances between all orally and intravenously administered fluids and all fluid losses
Blood coagulation markers | Up to the fifth postoperative day
  Parameters characterizing the humoral and cellular (thrombocytes) coagulation will be determined
Immunologic, endothelial and hepatic markers | Up to the fifth postoperative day
  Parameters characterizing the time course of immunological (e.g. Interleukin-6) and endothelial (e.g. Intercellular Adhesion Molecule 1) and hepatic (e.g. cytokeratin-18) response will be determined
Organ dysfunctions and complications | Up to the fifth postoperative day, at hospital discharge (an average of two weeks) and before, during and after the first cycle of chemotherapy (an average of four to six weeks)
  Organ complications are classified according to Clavien-Dindo classification
Microvascular function | Up to the fifth postoperative day and at hospital discharge (an average of two weeks)
  Microvascular function is assessed by near-infrared spectroscopy (NIRS) combined with a vascular occlusion test (VOT)
Functional status | At baseline, hospital discharge (expected average of 14 days) and before and after the first cycle of chemotherapy (an average of four to six weeks)
  Measured by the Barthel activities of daily living (ADL) index and activities of daily living (IADL)
Intensive care unit length of stay | Participants will be followed up until intensive care unit discharge (an average of two days)
  Time from admission to discharge from the intensive care unit
Hospital length of stay | Participants will be followed up until hospital discharge (expected average of 14 days)
  Time from admission to discharge from the hospital

OTHER OUTCOMES:
Quality of life | At baseline, hospital discharge (expected average of 14 days)
  Assessed with EQ-5D questionnaire by the EuroQol Group

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Hunsicker, MD, Principal Investigator — Department of Anesthesiology and Intensive Care Medicine, Campus Virchow Klinikum, Charité - University Medicine Berlin
Locations (1):
- Department of Anesthesiology and Intensive Care Medicine, Campus Charité Mitte and Campus Virchow Klinikum, Charité - University Medicine Berlin, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No